CLINICAL TRIAL: NCT03115931
Title: The Effect of Preoperative Nutritional Assessment and Nutritional Support on Clinical Outcomes in Elective Abdominal Surgery Patients: A Prospective Observational Study
Brief Title: The Effect of Preoperative Nutritional Assessment and Nutritional Support on Clinical Outcomes
Acronym: PNAS
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Collaborators: Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Xijing Hospital (Other); West China Hospital (Other); Xinqiao Hospital of Chongqing (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Changhai Hospital (Other); Shanghai 10th People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Wang Xinying, Professor, Chief of Clinical Nutrition Service, Jinling Hospital, China
Other Study IDs: 201502022-1
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Nutrition Assessment; Nutritional Support; Clinical Outcomes; General Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The serum were collected to assess the nutrition risk.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
It is a study to evaluate the relationship between preoperative nutritional assessment and clinical outcomes and to explore the effect of preoperative nutritional support on clinical outcomes in patients after abdominal operation.

DETAILED DESCRIPTION:
It is a multi-center prospective observational cohort study to evaluate the relationship between preoperative nutritional assessment and clinical outcomes and to explore the effect of preoperative nutritional support on clinical outcomes in patients after abdominal operation. The nutrition risk were evaluated by different methods. The nutrition support regimens and the clinical outcomes were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of patients or their legal representatives to participate in this study.
2. patients undergoing selective operation without trauma

Exclusion Criteria:

1. Age: <18 years old or >80 years old
2. Discharge within 24 hours
3. Accept surgery at 8:00 next day
4. Withdraw of patient's informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing selective operation without trauma.
Sampling Method: Probability Sample
Enrollment: 4880 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Morbidity of infection | From date of patients enrollment until the date of infection documented from any cause, assessed up to 2 months.
  Invasion of the host organism by microorganisms that can cause pathological conditions or diseases.

SECONDARY OUTCOMES:
Nutrition indicator | From date of patients enrollment until the date of patients discharge from hospital, assessed up to 2 months.
  albumin/prealbumin/transferrin/retinol binding protein/IL-6
Length of stay in hospital | From date of patients enrollment until the date of patients discharged from hospital, assessed up to 12 months.
  The length of patients stay in hospital.
Actual calories intake | From date of patients enrollment until the date of patients are subjected to operation, assessed up to 2 months.
  The total energy patients received during the study
Mortality | From date of patients enrollment until the date of death from any cause, assessed up to 2 months after patients discharged from hospital.
  All deaths reported in all enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, PhD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weimann A, Braga M, Harsanyi L, Laviano A, Ljungqvist O, Soeters P; DGEM (German Society for Nutritional Medicine); Jauch KW, Kemen M, Hiesmayr JM, Horbach T, Kuse ER, Vestweber KH; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Surgery including organ transplantation. Clin Nutr. 2006 Apr;25(2):224-44. doi: 10.1016/j.clnu.2006.01.015. Epub 2006 May 15. PMID 16698152
- [Background] Studley HO. Percentage of weight loss: a basic indicator of surgical risk in patients with chronic peptic ulcer. 1936. Nutr Hosp. 2001 Jul-Aug;16(4):141-3; discussion 140-1. No abstract available. PMID 11680474
- [Background] Wilmore DW, Dudrick SJ. Growth and development of an infant receiving all nutrients exclusively by vein. JAMA. 1968 Mar 4;203(10):860-4. No abstract available. PMID 4965871
- [Background] Braga M, Ljungqvist O, Soeters P, Fearon K, Weimann A, Bozzetti F; ESPEN. ESPEN Guidelines on Parenteral Nutrition: surgery. Clin Nutr. 2009 Aug;28(4):378-86. doi: 10.1016/j.clnu.2009.04.002. Epub 2009 May 21. PMID 19464088
- [Background] American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) Board of Directors. Clinical Guidelines for the Use of Parenteral and Enteral Nutrition in Adult and Pediatric Patients, 2009. JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):255-9. doi: 10.1177/0148607109333115. No abstract available. PMID 19398611
- [Background] Doig GS, Simpson F, Sweetman EA, Finfer SR, Cooper DJ, Heighes PT, Davies AR, O'Leary M, Solano T, Peake S; Early PN Investigators of the ANZICS Clinical Trials Group. Early parenteral nutrition in critically ill patients with short-term relative contraindications to early enteral nutrition: a randomized controlled trial. JAMA. 2013 May 22;309(20):2130-8. doi: 10.1001/jama.2013.5124. PMID 23689848